CLINICAL TRIAL: NCT02654028
Title: Association Between Autologous Transfusion and Recurrence-free Survival in Patients With Hepatocellular Carcinoma After Resection-a Prospective Non-randomized Controlled Trial
Brief Title: Association Between Autologous Transfusion and Recurrence-free Survival in Patients With HCC After Resection
Acronym: AT/HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Director, Guangxi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AT/HCC
Record Dates: First submitted 2016-01-10; First posted 2016-01-13 (Estimated); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Blood Transfusion, Autologous; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autotransfusion group (Experimental): These group of patients will receive autotransfusion before liver resection.
  Interventions: Procedure: Autotransfusion
- Control group (Active Comparator): These group of patients will not receive autotransfusion before liver resection.
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: Autotransfusion — These group of patients will receive autotransfusion before liver resection.
  Arms: Autotransfusion group
Other: Control group — These group of patients will not receive autotransfusion before liver resection.
  Arms: Control group

SUMMARY:
This prospective non-randomized controlled trial aims to determine whether autotransfusion of red blood cells salvaged before liver resection is associated with the recurrence-free survival in patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
Preoperative and intraoperative blood salvage autotransfusion is used in various surgical procedures. However, because of the risk of reinfusion of salvaged blood contaminated by tumor cells, the use of autotransfusion in hepatocellular carcinoma (HCC) patients undergoing liver resection is controversial. The critical points include whether tumor cells can be cleared by autotransfusion, whether autotransfusion increases the risk of recurrence or metastasis, and what are the indications for autotransfusion. Moreover, some other issues are still not addressed. For example, is it warranted to take the risk of tumor dissemination by using autotransfusion to avoid allogeneic blood transfusion? Do the remaining tumor cells after additional filtration by leukocyte depletion filters still possess potential tumorigenicity?

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent liver resection;
* Diagnosis of hepatocellular carcinoma confirmed by postoperative histopathology;
* Level of preoperative hemoglobin ≥110 g/L;
* Child-Pugh class A or B liver function;
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.

Exclusion Criteria:

* A history of other malignancies;
* History of active autoimmune or immunodeficiency diseases;
* Concurrent cardiac, pulmonary, cerebral, or renal dysfunction;
* Loss to follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with tumor recurrence | 1-year
  The 1-year tumor recurrence will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Hong Zhong, MD, Principal Investigator — Guangxi Medical University
Locations (1):
- Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi, China

REFERENCES:
- [Background] Han S, Kim G, Ko JS, Sinn DH, Yang JD, Joh JW, Lee SK, Gwak MS. Safety of the Use of Blood Salvage and Autotransfusion During Liver Transplantation for Hepatocellular Carcinoma. Ann Surg. 2016 Aug;264(2):339-43. doi: 10.1097/SLA.0000000000001486. PMID 26501715
- [Background] Tomimaru Y, Eguchi H, Wada H, Hama N, Kawamoto K, Kobayashi S, Umeshita K, Doki Y, Mori M, Nagano H. Predicting the necessity of autologous blood collection and storage before surgery for hepatocellular carcinoma. J Surg Oncol. 2013 Dec;108(7):486-91. doi: 10.1002/jso.23426. Epub 2013 Sep 5. PMID 24009154
- [Background] Kwon JH, Han S, Kim D, Kuk JH, Cho H, Kim S, Yang JD, Kim C, Kim JM, Choi GS, Joh JW, Ko JS, Gwak MS, Kim G. Blood Salvage and Autotransfusion With Single Leukoreduction Does Not Increase the Risk of Tumor Recurrence After Liver Transplantation for Advanced Hepatocellular Carcinoma. Ann Surg. 2022 Dec 1;276(6):e842-e850. doi: 10.1097/SLA.0000000000004866. Epub 2021 Mar 18. PMID 33914466